PROTOCOL TITLE: Administration Method of Cognitive Screening in Older Individuals With Hearing Loss

NCT#: 03402932

VERSION DATE: 11.25.2018

## Statistical analysis plan

The dependent variable is speech recognition outcome measure (MoCA test scores). The model include fixed effects of test modality (unamplified, amplified, visual), test version (A or B), and test period (1<sup>st</sup> or 2<sup>nd</sup>), as well as random by-participant intercept. The test modality condition is coded using simple coding strategy: the first contrast compares outcome measure between the unamplified and the amplified condition (-1/3, 2/3, -1/3); the second contrast compares outcome measure between the unamplified and the visual condition (-1/3, -1/3, 2/3). Both version and period are coded using simple coding as (-1/2, 1/2). Model are compared and selected based on AIC and Wald test results.